CLINICAL TRIAL: NCT04517630
Title: Acute Kidney Injury In Subjects With Severe Acute Respiratory Syndrome Due to SARS-CoV2 Infection
Brief Title: Renal Biomarkers in AKI and COVID-19
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Santiago Avila-Rios, Principal Investigator, Instituto Nacional de Enfermedades Respiratorias
Other Study IDs: C26-20
Record Dates: First submitted 2020-08-15; First posted 2020-08-18 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Coronavirus Infection; Covid19; SARS (Severe Acute Respiratory Syndrome); AKI
Keywords: AKI; SARS; METABOLOMIC; KIDNEY BIOMARKERS; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Severe Acute Respiratory Syndrome | interventions — Viral Load

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Biospecimen Retention: Samples With DNA — The SARS-CoV-2 RNA will be obtained from 200 microliters of urine, by standard methods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Severe pneumoniae: Evaluate the progression to AKI during first 30 days of recruitment
  Interventions: Diagnostic Test: urinary NGAL, TIMP-2, IGFBP7, IL-6, viral load and metabolomic

INTERVENTIONS:
Diagnostic Test: urinary NGAL, TIMP-2, IGFBP7, IL-6, viral load and metabolomic — Determine the evolution of NGAL, TIMP-2, IGFBP7, IL-6, viral load and metabolomic at basal, and the 3 , 5 and 7 days after recruitment

SUMMARY:
Severe pneumoniae related to Coronavirus Disease (COVID-19), had a high in-hospital mortality; this condition are worst in subjects with acute kidney disease (AKI); conditioning increased mortality, days of assisted mechanical ventilation (AMV), increased nosocomial infections and high costs. We need many studies for determinated the risk factors for AKI in subjects with COVID-19.

This study pretends identify the incidence of AKI in subjects with severe pneumoniae by COVID-19, describe the role of some biomarkers in the physiopathology of AKI-COVID-19; and determine the evolution of urinary biomarkers during hospitalization, like neutrophil gelatinase-associated lipocalin (NGAL), tissue inhibitor of metalloproteinases-2 (TIMP-2), insulin-like growth factor binding protein-7 (IGFBP7), and interleukin-6 (IL-6) and the progression of viruria of Severe Acute Respiratory Syndrome (SARS) related to CoronaVirus 2 (CoV2) in subjects with or without AKI.

DETAILED DESCRIPTION:
The usefulness of urinary NGAL levels and the platelet / lymphocyte index as predictive markers of AKI in the context of COVID-19 will be studied. These results will allow to propose more appropriate strategies for the prevention, diagnosis and timely management of patients with severe pneumonia due to COVID-19 and AKI. Knowing the viral load in urine and its evolution in patients with and without AKI will allow us to explore associations between the presence of the virus at the local level and the presence of kidney damage. Likewise, the presence of viral load in urine and its possible relationship with the local activation of the complement system, together with the detection of biomarkers of kidney damage, like NGAL, TIMP-2, IGFBP7, and IL-6, will allow us to better understand the pathophysiology of these alterations in the context of COVID-19; additionally, some patients received tocilizumab, an IL-6 inhibitor as a compassionate measure, which may reduce urinary levels of interleukins and other inflammatory markers.

Finally, the study of possible differences in the metabolome in urine in patients with and without acute kidney injury could favor the discovery of new markers to identify patients with SARS-CoV-2 infection susceptible to the development of AKI.

Determine the evolution of NGAL, TIMP-2, IGFBP7, IL-6, viral load and metabolomic basal, and the days 3 , 5 and 7 after recruitment

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age.
* Subjects admitted with a diagnosis of probable SARS-CoV-2 pneumonia.
* Subjects with a diagnosis of SARS-CoV-2 pneumonia confirmed by Real-time quantitative-Polymerase Chain Reaction (qRT-PCR).
* Subjects with qRT-PCR negative for SARS-CoV-2, but who meet clinical and radiological criteria for COVID-19, and no other causes have been identified.

Exclusion Criteria:

* Pregnant women
* Incomplete medical records.

Elimination criteria:

* Patients who die within the first 24 hours of entering the institute.
* Patients discharged for any reason not considered death within the first 48 hours, such as voluntary discharge or transfer to other health institutions.
* Patients who during their hospitalization report a positive PCR for other non-respiratory viruses without identifying SARS-CoV-2
* Patients who withdraw their consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Older adults were recruited, with a diagnosis of COVID-19 confirmed by PCR, in their first 48 hours of hospitalization that meet severity criteria, with 5 to 7 degrees of severity according to the WHO classification.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Urinary levels of renal biomarkers | Seven days
  To estimate the strength of association between the elevation of urinary levels of NGAL, TIMP-2, IGFBP7 and IL-6 and the development of AKI associated with SARS-CoV-2 pneumonia

SECONDARY OUTCOMES:
Incidence of AKI | One month
  Describe the incidence of AKI in critically ill patients with severe COVID-19 pneumonia
Urinary levels of renal biomarkers and mortality | 30 days
  Estimate the strength of association of elevated urinary levels of NGAL, TIMP-2, IGFBP7 and IL-6 with mortality
Urinary levels of renal biomarkers and severity of the disease. | 30 days
  Estimate the strength of association of elevated urinary levels of NGAL, TIMP-2, IGFBP7 and IL-6 with teh severity of the disease.
Risk factors for AKI in severe COVID-19 | 30 days
  Identify possible risk factors (epidemiological, clinical, paraclinical, use of nephrotoxic agents) for the development of AKI in critically ill patients with COVID-19 pneumonia.
Evolution renal biomarkers | 7 days
  Compare the evolution over time of renal function markers (NGAL, TIMP-2 and IGFBP7) in patients with and without kidney injury.
Evolution of viral load | 7 days
  Compare the evolution over time of the SARS-CoV-2 viral load in patients with and without acute kidney injury.
Evolution of complement pathway | seven days
  Analyze the complement pathway in urine and compare its evolution over time in patients with and without acute kidney injury and SARS-CoV-2 infection.
Metabolomic profile | 7 days
  Analyze the metabolomic profile in urine in patients with and without acute kidney injury with SARS-CoV-2 infection.
Respiratory changes | 30 days
  Describe partial arterial oxygen concentration/inspired oxygen faction (PaO2/FiO2) ratio and radiologic evolution in patients with severe SARS COV2 pneumonia.

OTHER OUTCOMES:
Nosocomial Infections | 30 days
  Stablish the nosocomial infections in subjects with or without AKI

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Avila Rios, PhD, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- Centro de Investigacion en Enfermedades Infecciosas, Mexico City, Mexico